CLINICAL TRIAL: NCT02367157
Title: Effectiveness of Kinesio Tape in Morning Stiffness and Functional Capacity in Patients With Rheumatoid Arthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEU-009
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Wrist Morning Stiffness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Kinesio taping (Experimental): Epicondilar and epitroclear muscle Kinesio Taping with a Space Correction on the wrist according Kenzo Kase Method
  Interventions: Procedure: Kenzo Kase Method; Device: Kinesio Taping
- No intervention: Control (No Intervention)

INTERVENTIONS:
Procedure: Kenzo Kase Method
  Arms: Experimental: Kinesio taping
Device: Kinesio Taping
  Arms: Experimental: Kinesio taping

SUMMARY:
The purpose of this study is to determine how the applications of Kinesio Tape affect the morning stiffness in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis according to the criteria of the American Rheumatism Association with a minimum of 6 months evolution from diagnosis.
* These subjects must have morning stiffness daily in the wrist joint of a member or bilateral at least a month.

Exclusion Criteria:

* Subjects in postoperative affecting the mobility of joints to study phase.
* Subjects with sensory deficits or other inflammatory arthropathies.
* Subjects who are or come in a state of emergence of the hand or wrist joints during the investigation.
* Subjects who change their usual treatment (medication or other therapies) two months before the study or during the study.
* We exclude subjects who present some kind of allergy to Kinesio-Tape in which case it will be removed immediately.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in the Wrist Morning Stiffness | participants will be followed for the duration in minutes of the morning stiffness, an expected average of 45 minutes]

CONTACTS AND LOCATIONS:
Locations (1):
- San Pablo CEU University, Boadilla del Monte, Madrid, Spain